CLINICAL TRIAL: NCT02146105
Title: A Yoga Exercise Intervention Designed for Women With Knee Osteoarthritis
Brief Title: Yoga as an Intervention for Women With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Yoga_KneeOA; Labarge (Other Grant/Funding Number: Labarge Optimal Aging Initiative)
Record Dates: First submitted 2014-05-16; First posted 2014-05-23 (Estimated); Results first posted 2015-02-19 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-08

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Yoga For Knee Osteoarthritis (Experimental): An tailored arthritis-specific yoga program for women with knee osteoarthritis with the aim of increasing leg strength and alleviating knee pain related to the disease.
  Interventions: Other: Yoga For Knee Osteoarthritis

INTERVENTIONS:
Other: Yoga For Knee Osteoarthritis — Yoga program specifically for women with knee osteoarthritis.

SUMMARY:
Keeping individuals with knee osteoarthritis physically active is critically important. Exercise is effective at reducing pain while improving physical function. However some exercises can overload the knee, and as a result, worsen knee pain and health of the knee joint. Yoga offers a foundation of static postures that improve muscle strength and joint flexibility. Using sophisticated technology that allows us to calculate the loads inside the knee, the investigators have selected yoga exercises that do not overload the knee joint. The investigators have designed a yoga exercise class that is ideal for people with knee osteoarthritis. The purpose of the study is to investigate whether these yoga exercises increase muscle strength and reduce knee pain in women with knee osteoarthritis. In addition, the investigators aim to show that these yoga exercises will also improve knee loads during activities, mobility and heart health. The investigators will ask 50 women with knee osteoarthritis to participate in a 12 week yoga exercise intervention, that requires attendance to 3 classes each week. The investigators will test strength of the leg muscles, pain, knee joint loads, mobility and cardiovascular health before and after the 12 week yoga exercise intervention.

DETAILED DESCRIPTION:
This study is an uncontrolled intervention study with repeated measures. The intervention is a 12-week supervised exercise class featuring biomechanically sound exercises for people with knee osteoarthritis. Measures of strength of the knee muscles, pain, biomechanics during walking and yoga, mobility and cardiovascular health will be included. Strength will be measured on a dynamometer. Pain will be assessed with questionnaires. Walking and three yoga postures will be observed using motion capture system integrated with force measurements from the floor. Mobility will be assessed during walking, stair-climbing and chair standing tasks. Cardiovascular health will be measured during a submaximal bicycle task.

ELIGIBILITY:
Inclusion Criteria:

* Female - 50 years of age or older
* Knee pain on most days of the week
* Less than 30 minutes of morning stiffness
* Bony enlargement
* Bony tenderness to palpation
* Signs of inflammation
* Able to safely climb 2 flights of stairs without aid
* Visited a family physician within the last 12 months

Exclusion Criteria:

* Any other forms of arthritis
* Osteoporosis
* History of patellofemoral symptoms
* Active non-arthritic knee disease
* Knee surgery
* Use of cane or walking aid
* Unstable heart condition
* Neurological conditions
* Skin allergy to medical tape
* Hip or ankle injuries in past 3 months
* Any injuries that would prohibit participation in yoga
* Ipsilateral hip or ankle conditions
* Currently receiving cancer treatment
* Currently pregnant

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica R Maly, PhD, Principal Investigator — School of Rehabilitation Sciences, McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Brenneman EC, Kuntz AB, Wiebenga EG, Maly MR. A Yoga Strengthening Program Designed to Minimize the Knee Adduction Moment for Women with Knee Osteoarthritis: A Proof-Of-Principle Cohort Study. PLoS One. 2015 Sep 14;10(9):e0136854. doi: 10.1371/journal.pone.0136854. eCollection 2015. PMID 26367862

RESULTS

PARTICIPANT FLOW:
Groups:
- Yoga Intervention: Participants completed a yoga strengthening program designed for knee osteoarthritis (OA). This program was taught by a certified yoga instructor who was trained to deliver the strengthening program. Participants were asked to attend 3 classes per week for 12 weeks. Each class was 1 hour in duration.
Period: Overall Study
Arm/Group | Yoga Intervention
Started | 45
Completed | 39
Not Completed | 6
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Arm/Group | Yoga For Knee Osteoarthritis
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Knee Extensor Torque
Description: Knee extensor torque (Newton*meter) is calculated on a Biodex dynamometer using an isometric protocol. Trials are completed as a voluntary maximum effort.
Time Frame: Week 1 and Week 13
Measure: Mean (Standard Deviation); unit: Nm
Arm/Group | Yoga For Knee Osteoarthritis
Number analyzed (Participants) | 45
Nm | 130.1 (42.1)

2. Primary Outcome: Change in Knee Pain
Description: Knee pain is assessed subjectively via the Knee Injury and Osteoarthritis Outcome Score (KOOS) and the Intermittent and Constant Osteoarthritis Pain (ICOAP) questionnaires.
Time Frame: Week 1 and Week 13
Reporting Status: Not Posted

3. Secondary Outcome: Change in Six Minute Walk Test (6MWT)
Description: Participants are asked to walk as far as possible for a total of six minutes at a self-selected pace in an obstruction-free rectangular hallway. Distance traveled is recorded in metres (m).
Time Frame: Week 1 and Week 13
Reporting Status: Not Posted

4. Secondary Outcome: Change in 30-second Chair Stand
Description: Participants are asked to cross their arms over their chest and rise and sit back down in a chair as many times as possible in 30 seconds.
Time Frame: Week 1 and Week 13
Reporting Status: Not Posted

5. Secondary Outcome: Change in Timed Up and Go (TUG)
Description: Participants are asked to raise from a standard chair, walk forward 3-metres until an orange cone is reached, walk around the cone, then walk back to the chair and sit down. The test is to be completed as quickly and safely as possible without running. The trial is repeated a second time and the quickest time (in seconds) is recorded.
Time Frame: Week 1 and Week 13
Reporting Status: Not Posted

6. Secondary Outcome: Change in Stair Ascent and Descent
Description: Participants are asked to climb a standard flight of 9 stairs as quickly and safely as possible without compromising safety. Stair ascent and descent are assessed individually. Time to climb the stairs are recorded (in seconds) and averaged over two trials.
Time Frame: Week 1 and Week 13
Reporting Status: Not Posted

7. Secondary Outcome: Change in Subjective Scales
Description: The Centre of Epidemiologic Studies Depression Scale (19-items), the Athens Insomnia Scale (8-items), and the Perceived Stress Scale (10-items) will be given to the participants to gather information on feelings of depression, sleeping patterns, and perceived stress, respectively.
Time Frame: Week 1 and Week 13
Reporting Status: Not Posted

8. Secondary Outcome: Change in Cardiovascular Fitness
Description: Cardiovascular fitness is assessed using a sub maximal oxygen consumption cycle ergometer test. Heart rate is monitored using a Polar Heart Rate monitor and the test is terminated upon one of two conditions: a) volitional fatigue, or b) within 10 beats of 85% of the age-predicted maximum heart rate is achieved. Values are recorded in mL/kg/min.
Time Frame: Week 1 and Week 13
Reporting Status: Not Posted

9. Secondary Outcome: Change in Biomechanical Outcomes
Description: Participants will be asked to partake in a complete kinematic, kinetic, and electromyographic analysis of gait and static postures using floor-embedded force plates, a 9-camera motion capture system, and a wireless electromyography system. Knee adduction moment (KAM; Nm/kg), normalized electromyography to a percentage of their maximal effort (%MVIC), and muscular co-activation (%) are the variables of interest.
Time Frame: Week 1 and Week 13
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Yoga For Knee Osteoarthritis
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 1/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Yoga For Knee Osteoarthritis (N=45)
Ankle injury (Musculoskeletal and connective tissue disorders) | 1 (1) — Painful ankle during the intervention period. Physician consultation revealed no fracture.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No